CLINICAL TRIAL: NCT02469675
Title: Paired Stimulation to Increase Cortical Transmission to Hand Muscles: Pilot Study
Brief Title: Brain and Nerve Stimulation for Hand Muscles in Spinal Cord Injury and ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Noam Y. Harel, MD, PhD, Staff Physician, Bronx VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HAR-15-001
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Spinal Cord Injury (SCI); Amyotrophic Lateral Sclerosis (ALS)
Keywords: Spinal Cord Injuries; Amyotrophic Lateral Sclerosis; Transcranial magnetic stimulation, single pulse; non-invasive brain stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Amyotrophic Lateral Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All subjects (Experimental): All subjects undergo same full protocol, including different combinations of stimulation on different days:
  Transcranial Magnetic Stimulation Cervical Transcutaneous Stimulation Median Nerve Stimulation
  Interventions: Device: Transcranial magnetic stimulation; Device: Median nerve stimulation; Device: Cervical transcutaneous stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — One TMS pulse every 10 seconds for 20 minutes
  Other Names: MagPro R30
Device: Median nerve stimulation — One median nerve pulse every 10 seconds for 20 minutes
  Other Names: Digitimer DS7A
Device: Cervical transcutaneous stimulation — One cervical pulse every 10 seconds for 20 minutes
  Other Names: Digitimer DS7A

SUMMARY:
Most neurological injuries such as spinal cord injuries (SCI) and amyotrophic lateral sclerosis (ALS) spare a portion of nerve circuitry. Strengthening spared nerve circuits may be an important method to improve functional recovery.

In this study, the investigators aim to use non-invasive magnetic and electrical stimulation to strengthen motor circuits between the brain and hands. Magnetic stimulation will be used over the motor cortex (scalp). Two methods of electrical stimulation will be compared: stimulation of the median nerve at the wrist; or direct stimulation of the cervical spinal cord across the skin on the back of the neck. Several different combinations of magnetic and electrical stimulation will be compared to find the conditions that best strengthen nerve circuits between the brain and hands - "Fire Together, Wire Together".

PLEASE NOTE, THIS IS A PRELIMINARY STUDY. This study is testing for temporary changes in nerve transmission and hand function. THERE IS NO EXPECTATION OF LONG-TERM BENEFIT FROM THIS STUDY. If we see temporary changes in this study, then future studies would focus on how to prolong that effect.

DETAILED DESCRIPTION:
Most neurological injuries such as spinal cord injuries (SCI) and amyotrophic lateral sclerosis (ALS) spare a portion of nerve circuitry. Strengthening spared nerve circuits represents a critical method to improve functional recovery. Different forms of magnetic and electrical stimulation have been used to activate brain, spinal cord, nerve, or muscle tissue. Although in some cases, surgically implanted electrical stimulation has delivered tremendous benefit, a non-invasive approach to nerve stimulation is preferable.

In this proposed study, the investigators aim to use non-invasive magnetic and electrical stimulation to strengthen motor circuits between the brain and hands. Transcranial magnetic stimulation (TMS) will be combined with either electrical stimulation of the median nerve at the wrist; or electrical transcutaneous stimulation of the cervical spinal cord. Magnetic and electrical stimulation will be precisely timed so that the pulses arrive at the target spinal motor neurons at roughly the same time - this precise timing is responsible for the phenomenon of "spike timing-dependent plasticity".

Three groups of participants will be studied: individuals with chronic incomplete cervical SCI (n=12), individuals with definite or probable ALS (n=6), and individuals without neurological injury or disease (n=12). Subjects with SCI or ALS will have one screening visit to confirm eligibility for the study. All subjects will then undergo one baseline testing session followed by 7 sessions of unpaired or paired magnetic and electrical stimulation. Functional and physiological testing will be conducted prior to each stimulation session, then at 0, 15, 30, and 90 minutes post each session. Key measures include grip strength dynamometry, timed performance on a hand dexterity test, amplitude of abductor pollicis brevis (APB) response to TMS, integrated amplitude of APB F-wave responses, and duration of the 'cortical silent period' after TMS stimulation during APB contraction.

PLEASE NOTE, THIS IS A PRELIMINARY STUDY. This study is testing for temporary changes in nerve transmission and hand function. THERE IS NO EXPECTATION OF LONG-TERM BENEFIT FROM THIS STUDY. If we see temporary changes in this study, then future studies would focus on how to prolong that effect.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 21-65 years;
* No history of serious neurological injury or disease; OR
* Chronic (>12 months since injury) incomplete SCI between levels C2-C8 or diagnosis of definite or probable ALS;
* Incomplete weakness of left or right hand muscles: score of 3 or 4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction;
* Detectable F-wave responses of the left or right abductor pollicis brevis muscle to median nerve stimulation;
* Detectable motor evoked potentials in left or right abductor pollicis brevis muscle to transcranial magnetic stimulation.

Exclusion Criteria:

* Multiple spinal cord lesions;
* History of seizures;
* Ventilator dependence or patent tracheostomy site;
* Use of medications that significantly lower seizure threshold, such as tricyclic antidepressants, amphetamines, neuroleptics, dalfampridine, and bupropion;
* History of stroke, brain tumor, brain abscess, or multiple sclerosis;
* History of moderate to severe head trauma (loss of consciousness for greater than one hour or evidence of brain contusion or hemorrhage or depressed skull fracture on prior imaging);
* History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants, or cardiac pacemaker/defibrillator;
* Significant coronary artery or cardiac conduction disease;
* Recurrent history over the last 6 months of autonomic dysreflexia;
* History of bipolar disorder;
* History of suicide attempt;
* Active psychosis;
* Heavy alcohol consumption (greater than equivalent of 5 oz of liquor) within previous 48 hours;
* Open skin lesions over the face, neck, shoulders, or arms;
* Pregnancy;
* Unsuitable for study participation as determined by study physician.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-06; Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in motor evoked potential (MEP) amplitude of the abductor pollicis brevis (APB) muscle response to single pulses of TMS | Assessed pre, then 0, 15, 30, and 90 minutes post-intervention.
Hand dexterity | Assessed pre, then 0, 15, 30, and 90 minutes post-intervention.
  Timed performance on a grooved pegboard task.
Safety and tolerability | Assessed periodically during each session.
  Vital signs are monitored throughout procedure; symptoms and degree of pain/discomfort are checked frequently.

SECONDARY OUTCOMES:
Grip strength | Assessed pre, then 0, 15, 30, and 90 minutes post-intervention.
  Strength will be quantified using hand-held wireless dynamometry.
Change in the duration of the 'cortical silent period' after TMS stimulation during APB contraction | Assessed pre, then 0, 15, 30, and 90 minutes post-intervention.
F-wave responses of the APB muscle | Assessed pre, then 0, 15, 30, and 90 minutes post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y. Harel, MD, PhD, Principal Investigator — James J. Peters VA Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
A Limited Dataset (LDS) will be shared in electronic format pursuant to a VA-approved Data Use Agreement. Individually Identifiable Data will be shared pursuant to valid HIPAA Authorization, Informed Consent, and an appropriate written agreement limiting use of the data to the conditions as described in the authorization and consent, and a written assurance from the recipient that the information will be maintained in accordance with the security requirements of 38 CFR Part 1.466.